CLINICAL TRIAL: NCT05587543
Title: Clinical Study on the Safety and Efficacy of EBV CAR-T /TCR-T Cells in the Treatment of Recurrent / Refractory EBV Positive Nasopharyngeal Carcinoma
Brief Title: Clinical Study on the EBV CAR-T /TCR-T Cells in the Treatment of Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Chief Doctor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2207257-17
Record Dates: First submitted 2022-09-27; First posted 2022-10-20 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Automobiles; Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: CAR-T、TCR-T
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAR-T (Experimental): Target A positivity was assigned to CAR-T cell therapy.
  Interventions: Behavioral: PK Blood Collection; Drug: CAR
- TCR-T (Experimental): Target A negative, Target B positive and Target C positive were assigned to TCR-T cell treatment group.
  Interventions: Behavioral: PK Blood Collection; Drug: TCR

INTERVENTIONS:
Behavioral: PK Blood Collection — All subjects were subjected to PK blood sampling as prescribed by the protocol.
Drug: CAR — Target A positive subjects will receive CAR-T cell therapy.
  Other Names: CAR-T cell therapy
  Arms: CAR-T
Drug: TCR — Target A negative, Target B positive and Target C positive subjects will receive TCR-T cell therapy.
  Other Names: TCR -T cell therapy
  Arms: TCR-T

SUMMARY:
This study was a single-arm, open-label, "3 + 3" dose-escalation Exploratory research. The patients were divided into two groups: EBV TCR-T-cell Group and EBV CAR-T-cell group. The EBV CAR-T-treated group received three progressively increasing dose levels (3.0 × 106 cells/kg, 9.0 × 106 cells/kg, 1.5 × 107 cells/kg) of EBV CAR-T-cell therapy; The EBV TCR-T-cell group received three progressively increasing doses (5.0 × 106 cells/kg, 1.5 × 107 cells/kg, 3.0 × 107 cells/kg) of EBV TCR-T-cell therapy.

DETAILED DESCRIPTION:
Each subject was observed for at least 4 weeks after cell reinfusion (DLT observation period) . A minimum of three participants should be included in each dose group, and two or more participants should not be included in each dose group at the same time, each subject should not be enrolled until the first 1 subject did not experience a grade 3 or higher adverse event (CTCAE5.0) related to the study drug during the DLT observation period. Three or six subjects were enrolled in each dose group, depending on the occurrence of DLT. If three subjects in one dose group did not experience DLT, three subjects were enrolled in the next higher dose group; if one of three subjects experienced DLT, three more subjects were enrolled in the dose group; Expanded to 6 subjects; if only 1 of the 6 subjects after amplification produced a DLT, then 3 subjects were enrolled into the next higher dose; If a DLT occurred in ≥2 of the 6 subjects after amplification, then the dose was specified to be higher than the MTD (MTD defined as the highest dose at which a DLT occurred in ≤1/6 subjects) , new subjects were included in the previous lower dose (tolerated dose) group until the lower dose group reached 6 subjects. If DLT occurred in ≤1/6 of the subjects, the lower dose group was defined as MTD or the best effective dose. A total of six subjects received the maximum tolerated dose. In the course of the study, the researcher can combine the safety and preliminary efficacy data of the enrolled subjects, and take the safety of the subjects and the maximum benefit of the disease as the premise, study treatment was performed at the maximum tolerated dose or other doses determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent;
* Age ≥18 years old, ≤75 years old, male and female;
* Expected survival ≥3 months;
* The Eastern Cooperative Oncology Group (ECOG) physical fitness score was 0-2;
* Ebv-positive nasopharyngeal carcinoma was diagnosed by in situ hybridization with Ebers (Eber-fish) .
* Pathological Paraffin section testing (within 5 years before signing the informed consent form) ;
* At least one measurable lesion according to RECIST v1.1 criteria for solid tumors;
* Recurrent/metastatic nasopharyngeal carcinoma patients who had previously failed second-line or more systemic therapy;
* An apheresis or venous access can be established and there are no other contraindications to blood cell isolation；
* CTCAE 5.0 was lower than grade 1 in the side effects of previous anti-tumor therapy (radiotherapy, chemotherapy, targeted therapy, etc.)
* During the study period and up to 6 months after the end of the administration, fertile subjects -LRB-both male and female) were required to use effective medical contraception. For women of reproductive age, a pregnancy test should be performed within 72 hours before the first dose, and the results were negative.

Exclusion Criteria:

* Active central nervous system metastases (except those that are stable after treatment)；
* HIV positive, HBsAg positive and HBV DNA copy number positive (quantitative detection ≥1000 CPS/ml) , HCV antibody positive and HCV RNA positive;
* Patients with mental or psychological disorders who can not cooperate with the treatment and evaluation of the curative effect;
* Subjects with severe autoimmune disease and long-term use of immunosuppressants;
* Active or uncontrolled infection requiring systemic therapy was present within 14 days prior to enrollment；
* Any unstable systemic disease;
* Complicated with dysfunction of important organs such as lung, brain and kidney.
* Subjects had undergone major surgery or severe trauma within 4 weeks before receiving cell therapy, or were expected to undergo major surgery during the study period.
* Participants received their last dose of radiation or anti-tumor therapy within 4 weeks of receiving the cell therapy.
* Participants had or had had other cancers that were incurable for up to 3 years, except for cervical cancer in situ or skin basal-cell carcinoma, and other cancers that had disease-free survival of more than 5 years.
* Treated with Chimeric antigen receptor t-cell therapy within six months.
* Graft-versus-host disease (GVHD)；
* Subjects who were receiving systemic steroid therapy before screening and who required long-term systemic steroid therapy during treatment as determined by the investigator (with the exception of inhaled or topical use) ; And subjects treated with systemic steroids within 72 hours before cell reinfusion (except for inhalation or topical use) .
* Severe allergies or a history of allergies;
* Subjects requiring anticoagulant therapy;
* Pregnant or lactating women, or a six-month pregnancy plan (for both men and women)；
* Researchers believe there are other reasons not to include people in treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | one year
  Analysis based on clinical trial data of subjects
MTD or the best effective dose | one year
  Analysis based on clinical trial data of subjects
Incidence of AE、SAE、AESI | one year
  Analysis based on clinical trial data of subjects

SECONDARY OUTCOMES:
PK parameter：Cmax | one year
  Analysis based on clinical trial data of subjects
PK parameter：Tmax | one year
  Analysis based on clinical trial data of subjects
ORR | one year
  Analysis based on clinical trial data of subjects
DCR | one year
  Analysis based on clinical trial data of subjects
DOR | one year
  Analysis based on clinical trial data of subjects
PFS | one year
  Analysis based on clinical trial data of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, Doctorate, Principal Investigator — Fudan University
Locations (1):
- Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taylor GS, Long HM, Brooks JM, Rickinson AB, Hislop AD. The immunology of Epstein-Barr virus-induced disease. Annu Rev Immunol. 2015;33:787-821. doi: 10.1146/annurev-immunol-032414-112326. Epub 2015 Feb 11. PMID 25706097
- [Result] Dalton T, Doubrovina E, Pankov D, Reynolds R, Scholze H, Selvakumar A, Vizconde T, Savalia B, Dyomin V, Weigel C, Oakes CC, Alonso A, Elemento O, Pan H, Phillip JM, O'Reilly RJ, Gewurz BE, Cesarman E, Giulino-Roth L. Epigenetic reprogramming sensitizes immunologically silent EBV+ lymphomas to virus-directed immunotherapy. Blood. 2020 May 21;135(21):1870-1881. doi: 10.1182/blood.2019004126. PMID 32157281
- [Result] Castillo JJ, Beltran BE, Miranda RN, Paydas S, Winer ES, Butera JN. Epstein-barr virus-positive diffuse large B-cell lymphoma of the elderly: what we know so far. Oncologist. 2011;16(1):87-96. doi: 10.1634/theoncologist.2010-0213. Epub 2011 Jan 6. PMID 21212426
- [Result] Dojcinov SD, Fend F, Quintanilla-Martinez L. EBV-Positive Lymphoproliferations of B- T- and NK-Cell Derivation in Non-Immunocompromised Hosts. Pathogens. 2018 Mar 7;7(1):28. doi: 10.3390/pathogens7010028. PMID 29518976
- [Result] Thompson MP, Kurzrock R. Epstein-Barr virus and cancer. Clin Cancer Res. 2004 Feb 1;10(3):803-21. doi: 10.1158/1078-0432.ccr-0670-3. PMID 14871955
- [Result] Kimura H, Fujiwara S. Overview of EBV-Associated T/NK-Cell Lymphoproliferative Diseases. Front Pediatr. 2019 Jan 4;6:417. doi: 10.3389/fped.2018.00417. eCollection 2018. PMID 30662890
- [Result] Healy JA, Dave SS. The Role of EBV in the Pathogenesis of Diffuse Large B Cell Lymphoma. Curr Top Microbiol Immunol. 2015;390(Pt 1):315-37. doi: 10.1007/978-3-319-22822-8_13. PMID 26424652
- [Result] Mao Y, Zhang DW, Zhu H, Lin H, Xiong L, Cao Q, Liu Y, Li QD, Xu JR, Xu LF, Chen RJ. LMP1 and LMP2A are potential prognostic markers of extranodal NK/T-cell lymphoma, nasal type (ENKTL). Diagn Pathol. 2012 Dec 13;7:178. doi: 10.1186/1746-1596-7-178. PMID 23237707
- [Result] Wang ZY, Liu QF, Wang H, Jin J, Wang WH, Wang SL, Song YW, Liu YP, Fang H, Ren H, Wu RY, Chen B, Zhang XM, Lu NN, Zhou LQ, Li YX. Clinical implications of plasma Epstein-Barr virus DNA in early-stage extranodal nasal-type NK/T-cell lymphoma patients receiving primary radiotherapy. Blood. 2012 Sep 6;120(10):2003-10. doi: 10.1182/blood-2012-06-435024. Epub 2012 Jul 23. PMID 22826562
- [Result] Cho SG, Kim N, Sohn HJ, Lee SK, Oh ST, Lee HJ, Cho HI, Yim HW, Jung SE, Park G, Oh JH, Choi BO, Kim SW, Kim SW, Chung NG, Lee JW, Hong YS, Kim TG. Long-term Outcome of Extranodal NK/T Cell Lymphoma Patients Treated With Postremission Therapy Using EBV LMP1 and LMP2a-specific CTLs. Mol Ther. 2015 Aug;23(8):1401-1409. doi: 10.1038/mt.2015.91. Epub 2015 May 28. PMID 26017177
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Chen YP, Chan ATC, Le QT, Blanchard P, Sun Y, Ma J. Nasopharyngeal carcinoma. Lancet. 2019 Jul 6;394(10192):64-80. doi: 10.1016/S0140-6736(19)30956-0. Epub 2019 Jun 6. PMID 31178151
- [Result] Wang L, Tian WD, Xu X, Nie B, Lu J, Liu X, Zhang B, Dong Q, Sunwoo JB, Li G, Li XP. Epstein-Barr virus nuclear antigen 1 (EBNA1) protein induction of epithelial-mesenchymal transition in nasopharyngeal carcinoma cells. Cancer. 2014 Feb 1;120(3):363-72. doi: 10.1002/cncr.28418. Epub 2013 Nov 4. PMID 24190575
- [Result] Zhu S, Chen J, Xiong Y, Kamara S, Gu M, Tang W, Chen S, Dong H, Xue X, Zheng ZM, Zhang L. Novel EBV LMP-2-affibody and affitoxin in molecular imaging and targeted therapy of nasopharyngeal carcinoma. PLoS Pathog. 2020 Jan 6;16(1):e1008223. doi: 10.1371/journal.ppat.1008223. eCollection 2020 Jan. PMID 31905218
- [Result] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Result] Lee AW, Ng WT, Chan LL, Hung WM, Chan CC, Sze HC, Chan OS, Chang AT, Yeung RM. Evolution of treatment for nasopharyngeal cancer--success and setback in the intensity-modulated radiotherapy era. Radiother Oncol. 2014 Mar;110(3):377-84. doi: 10.1016/j.radonc.2014.02.003. Epub 2014 Mar 11. PMID 24630534
- [Result] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Result] Oliva M, Huang SH, Taylor R, Su J, Xu W, Hansen AR, Jang R, Bayley A, Hosni A, Giuliani M, Ringash J, Bratman SV, Cho J, Irish J, Waldron J, Weinreb I, Kim J, O'Sullivan B, Siu LL, Spreafico A. Impact of cumulative cisplatin dose and adjuvant chemotherapy in locally-advanced nasopharyngeal carcinoma treated with definitive chemoradiotherapy. Oral Oncol. 2020 Jun;105:104666. doi: 10.1016/j.oraloncology.2020.104666. Epub 2020 Apr 6. PMID 32272384
- [Result] Zhang E, Gu J, Xu H. Prospects for chimeric antigen receptor-modified T cell therapy for solid tumors. Mol Cancer. 2018 Jan 12;17(1):7. doi: 10.1186/s12943-018-0759-3. PMID 29329591
- [Result] Castellarin M, Watanabe K, June CH, Kloss CC, Posey AD Jr. Driving cars to the clinic for solid tumors. Gene Ther. 2018 Jun;25(3):165-175. doi: 10.1038/s41434-018-0007-x. Epub 2018 Jun 7. PMID 29880908